CLINICAL TRIAL: NCT02450942
Title: Radiation Dosimetry, Plasma Pharmacokinetics, Biodistribution, Safety and Diagnostic Performance of 18F-FDS PET/CT in Healthy Volunteers and Patients With Suspected Infection
Brief Title: 18F-FDS PET/CT in Healthy Volunteers and Patients With Suspected Infection
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PUMCHNM08
Record Dates: First submitted 2015-05-13; First posted 2015-05-21 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2015-05

CONDITIONS: Enterobacteriaceae Infections
MeSH Terms: conditions — Enterobacteriaceae Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 18F-FDS injection and PET/CT scan (Experimental): The patients were intravenously injected with 18F-FDS and underwent PET/CT scan 1 h after the injection.
  Interventions: Drug: 18F-FDS

INTERVENTIONS:
Drug: 18F-FDS — 18F-FDS were intravenously injected into the patients 1 h before the PET/CT scans
  Other Names: 2-[18F]-fluorodeoxysorbitol

SUMMARY:
This is an open-label dynamic whole-body PET/CT (positron emission tomography/computed tomography) study for investigation of radiation dosimetry, plasma pharmacokinetics, biodistribution, safety and diagnostic performance of 18F-FDS in healthy volunteers and patients with suspected infection. A single dose of nearly 370 MBq 18F-FDS will be intravenously injected into healthy volunteers and patients with suspected infection. Visual and semiquantitative method will be used to assess the PET/CT images. Changes of blood pressure, pulse, respiration, temperature, routine blood and urine tests, serum alanine aminotransferase, albumin, and creatinine, and any adverse events will be collected from the volunteers. Adverse events will also be observed in the patients.

DETAILED DESCRIPTION:
In clinical microbiology, pathogenic enterobacteriaceae are differentiated from other organisms by selectively metabolizing sorbitol. They exclusively express the enzyme sorbitol-6-phosphate dehydrogenase, which is the enzyme responsible for initiating sorbitol metabolism. 2-[18F]-fluorodeoxysorbitol (18F-FDS) is a positron-emitting analog of sorbitol. The substitution of the hydroxyl group by fluorine at the C-2 position, however, completely abrogates the recognition by mammalian sorbitol dehydrogenase.18F-FDS could be a suitable probe to selectively label and tomographically image enterobacteriaceae in vivo.

For further interests in clinical translation of 18F-FDS, an open-label dynamic whole-body PET/CT study was designed to investigate radiation dosimetry, plasma pharmacokinetics, biodistribution, safety and diagnostic performance of 18F-FDS in healthy volunteers and patients with suspected infection. A single dose of nearly 370 MBq 18F-FDS will be intravenously injected into healthy volunteers and patients with suspected infection. Visual and semiquantitative method will be used to assess the PET/CT images. Changes of blood pressure, pulse, respiration, temperature, routine blood and urine tests, serum alanine aminotransferase, albumin, and creatinine, and any adverse events will be collected from the volunteers. Adverse events will also be observed in the patients.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers:

  o Males and females, ≥18 years old
* Infectious patients:

  * Males and females, ≥18 years old
  * Characteristic clinical signs, symptoms and laboratory tests suggesting the diagnosis of infectious disease.
  * The diagnosis of infection is based on The Centres for Disease Control and Prevention (CDC) criteria for diagnosing infection. They rely on a combination of clinical, radiological, operative, microbiological, and histological findings, in addition to results of other laboratory tests, such as the white blood cell count, erythrocyte sedimentation rate, and C reactive protein value.

Exclusion Criteria:

* Females planning to bear a child recently or with childbearing potential
* Renal function: serum creatinine >3.0 mg/dL (270 μM/L)
* Liver function: any hepatic enzyme level more than 5 times upper limit of normal.
* Known severe allergy or hypersensitivity to IV radiographic contrast.
* Patients not able to enter the bore of the PET/CT scanner.
* Inability to lie still for the entire imaging time because of cough, pain, etc.
* Inability to complete the needed examinations due to severe claustrophobia, radiation phobia, etc.
* Concurrent severe and/or uncontrolled and/or unstable other medical disease that, in the opinion of the Investigator, may significantly interfere with study compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-01; Primary Completion 2018-01 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Visual and semiquantitative assessment of lesions and biodistribution | One year
  Visual analysis will be performed by consensus reading by at least 3 experienced nuclear medicine physician. The semiquantitative analysis will be performed by the same person for all the cases, and the standardized uptake values (SUVs) of tumor and organs will be measured.

SECONDARY OUTCOMES:
Blood pressure | 24 hours
  Blood pressure of healthy volunteers will be measured at three time points: right before injection, after scanning, and 24 hours after treatment.
Pulse | 24 hours
  Pulse will be measured at three time points for each healthy volunteer: right before injection, after scanning, and 24 hours after treatment.
Respiration frequency | 24 hours
  Respiration frequency will be measured at three time points for each healthy volunteer: right before injection, after scanning, and 24 hours after treatment.
Temperature | 24 hours
  Temperature will be measured at three time points for each healthy volunteer: right before injection, after scanning, and 24 hours after treatment.
Routine blood test | 24 hours
  Routine blood test of healthy volunteers will be measured at two time points: right before injection and 24 hours after treatment.
Routine urine test | 24 hours
  Routine urine test of healthy volunteers will be measured at two time points: right before injection and 24 hours after treatment.
Serum alanine aminotransferase | 24 hours
  Serum alanine aminotransferase of healthy volunteers will be measured at two time points: right before injection and 24 hours after treatment.
Serum albumin | 24 hours
  Serum albumin of healthy volunteers will be measured at two time points: right before injection and 24 hours after treatment.
Serum creatinine | 24 hours
  Serum creatinine of healthy volunteers will be measured at two time points: right before injection and 24 hours after treatment.
Adverse events collection | 5 days
  Adverse events within 5 days after the injection and scanning of healthy volunteers and patients will be followed and assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaohui Zhu, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kong Z, Wang Y, Ma W, Cheng X. Role of 18F-fluorodeoxyglucose (FDG) and 18F-2-fluorodeoxy sorbitol (FDS) in autoimmune hypophysitis: a case report. BMC Endocr Disord. 2020 Jun 9;20(1):84. doi: 10.1186/s12902-020-00567-8. PMID 32517690
- [Derived] Yao S, Xing H, Zhu W, Wu Z, Zhang Y, Ma Y, Liu Y, Huo L, Zhu Z, Li Z, Li F. Infection Imaging With (18)F-FDS and First-in-Human Evaluation. Nucl Med Biol. 2016 Mar;43(3):206-14. doi: 10.1016/j.nucmedbio.2015.11.008. Epub 2015 Dec 4. PMID 26924501